CLINICAL TRIAL: NCT04457245
Title: Phase 3 Randomized Trial Of PSMA PET Prior to Definitive Radiation Therapy for Unfavorable Intermediate-Risk or High-Risk Prostate Cancer [PSMA dRT]
Brief Title: Randomized Trial of PSMA PET Scan Before Definitive Radiation Therapy for Prostate Cancer
Acronym: PSMA-dRT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-000378; NCI-2020-03445 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Stage I Prostate Cancer American Joint Committee on Cancer (AJCC) v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
Keywords: PSMA; PET/CT; randomized trial; definitive Radiation Therapy; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (dRT) (Active Comparator): 150 Patients undergo standard dRT at the discretion of the treating radiation oncologist. Patient does not undergo PSMA PET for RT planning. Any other imaging is allowed, including CT/BS/MR/PET depending on local practice. No other primary treatment can be given before dRT. If a patient assigned to the control arm undergo a PSMA PET scan at another institution he will be discontinued from the study.
  Interventions: Radiation: Radiation Therapy
- Arm II (18F-DCFPyL, PET/CT, dRT) (Experimental): 162 Patient undergoes PSMA PET with 18F-DCFPyL for dRT planning. Any other imaging is allowed, including CT/BS/MR/PET depending on local practice. Patients then undergo dRT at the discretion of the treating radiation oncologist, who receives PSMA PET results and images. No other primary treatment can be given before RT.
  Interventions: Procedure: Computed Tomography; Other: Fluorine F 18 DCFPyL; Procedure: Positron Emission Tomography; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Computed Tomography — Undergo whole body PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
  Arms: Arm II (18F-DCFPyL, PET/CT, dRT)
Other: Fluorine F 18 DCFPyL — Given IV
  Other Names: 18F-DCFPyL
  Arms: Arm II (18F-DCFPyL, PET/CT, dRT)
Procedure: Positron Emission Tomography — Undergo whole body PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
  Arms: Arm II (18F-DCFPyL, PET/CT, dRT)
Radiation: Radiation Therapy — Undergo standard of care definitive radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This randomized phase III trial studies the success rate of definitive radiation therapy (dRT) for prostate cancer (PCa) with or without planning based on PSMA PET. PSMA- PET-based dRT, may improve radiation therapy planning and patient selection for dRT, and potentially improve its outcome compared to dRT without PSMA PET (standard dRT).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the outcome of patients with unfavorable intermediate (IR) and high-risk (HR) prostate cancer (PCa) after standard dRT versus prostate-specific membrane antigen (PSMA) positron emission tomography (PET)-based dRT.

OUTLINE: Patients are randomized to 1 of 2 arms. In both arms, no other primary treatment should be given before RT.

Arm I: Patients do not undergo PSMA PET for dRT planning. Patients undergo standard of care dRT at the discretion of the treating radiation oncologist.

Arm II: Patients undergo PSMA PET for dRT planning. Patients then undergo dRT at the discretion of the treating radiation oncologist, who receives the PSMA PET result and images.

After completion of dRT, clinical follow-up of patients with their treating radiation oncologist will be obtained for 5 years. The investigators will rely on the medical records obtained from the treating physicians as the primary source of outcome data.

ELIGIBILITY:
Inclusion Criteria:

* Adult male 18 years or older
* Histopathologically-proven PCa
* Unfavorable IR to HR disease:

  * Prostate specific antigen (PSA) >= 10 ng/mL
  * Or cT-stage >= 2b
  * Or Gleason grade 3 (4+3=7) or higher
  * Or Gleason grade 2 (3+4=7) AND >= 50% positive biopsy cores
  * Or Decipher Score >= 0.45
* Treating radiation oncologist intends to incorporate PSMA PET findings into the radiotherapy plan, if patient undergoes PSMA PET (intervention arm 2)
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Less than 18 years old at the time of investigational product administration
* Extra-pelvic metastasis (M1 disease) on any imaging or biopsy done before randomization
* Prior PSMA PET
* Prior pelvic RT
* Contraindications to radiotherapy (including active inflammatory bowel disease)
* Concurrent or prior surgery or systemic therapy for PCa at the time of randomization

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Success rate of definitive radiation therapy (dRT) | From date of randomization to first occurrence of progression, assessed up to 5 years
  Will be measured as progression-free survival after initiation of dRT. Progression is defined as (whichever occurs first): A biochemical recurrence defined as a rise by 2 ng/mL or more above the nadir prostate specific antigen (PSA) (defined as the lowest PSA achieved) after radiotherapy with or without short-term hormonal therapy, appearance of metastasis or loco-regional recurrence (diagnosed by any imaging or biopsy), initiation of any new salvage therapy or death from any cause. Survival curves will be constructed using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Loco-regional progression free survival | Up to 5 years after the date of randomization
  Diagnosis of local recurrence or pelvic nodal disease (N1) can be obtained by any imaging or biopsy.
Metastasis-free survival after initiation of radiation therapy (RT) | Up to 5 years after the date of randomization
  Diagnosis of extra-pelvic metastatic (M1) disease can be obtained by any imaging or biopsy.
Overall survival | Up to 5 years after the date of randomization
Change in initial treatment intent | Baseline up to 5 years after the date of randomization
  Will estimate the proportion of subjects in the prostate-specific membrane antigen (PSMA) group that have a change in the initial treatment intent and compute a 95% confidence interval for that proportion.
PSMA positron emission tomography (PET) derived predictors of progression-free survival | Up to 5 years after the date of randomization
  Will use Cox-proportional hazards regression to assess PSMA PET predictors of progression-free survival.
PSMA PET derived predictors of overall survival | Up to 5 years after the date of randomization
  Will use Cox-proportional hazards regression to assess PSMA PET predictors of overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Calais J, Zhu S, Hirmas N, Eiber M, Hadaschik B, Stuschke M, Herrmann K, Czernin J, Kishan AU, Nickols NG, Elashoff D, Fendler WP. Phase 3 multicenter randomized trial of PSMA PET/CT prior to definitive radiation therapy for unfavorable intermediate-risk or high-risk prostate cancer [PSMA dRT]: study protocol. BMC Cancer. 2021 May 7;21(1):512. doi: 10.1186/s12885-021-08026-w. PMID 33962579